CLINICAL TRIAL: NCT07305714
Title: Virtual Reality Educational Intervention for Nursing Students' Day Surgery Patient Counselling: A Mixed-Methods Pilot Feasibility Study
Brief Title: Virtual Reality Educational Intervention for Nursing Students' Day Surgery Patient Counselling
Acronym: CINDY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seinajoki University of Applied Sciences (Other)
Collaborators: Tampere University (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Terhi Voltti, Doctoral Candidate, Lecturer, MSc, Seinajoki University of Applied Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CINDY-2025-SEAMK; Ethics-20251108 (Other: Seinäjoki University of Applied Sciences)
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Virtual Reality; Nursing Education; Ambulatory Surgery; Day Surgery; Patient Counselling; Patient Education; Nursing Students; Perioperative Nursing; Feasibility Studies; Mixed Methods Studies

STUDY DESIGN:
Intervention Model Description: Non-randomized parallel group design with intervention group (n=30) receiving CINDY VR intervention plus standard education and control group (n=30) receiving standard education only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Nursing students (n=30) receive the CINDY virtual reality educational intervention (90 minutes, ThingLink platform) in addition to standard perioperative nursing education. The VR intervention includes interactive 360-degree scenarios showing day surgery patient journeys from the patient's perspective.
  Interventions: Behavioral: CINDY Virtual Reality Educational Intervention
- Control Group (No Intervention): Nursing students (n=30) receive standard perioperative nursing education only, without the CINDY VR intervention.

INTERVENTIONS:
Behavioral: CINDY Virtual Reality Educational Intervention — The CINDY (Counseling Intervention for Day Surgery) is a 90-minute virtual reality-based educational program delivered through the ThingLink platform. The intervention features interactive 360-degree VR scenarios depicting day surgery patient journeys from admission through discharge, including preoperative preparation, postoperative recovery, and discharge counseling. The scenarios were co-designed by a nursing educator, digital content expert, and day surgery nurse, and filmed in authentic clinical settings. Students experience situations from the patient's perspective, focusing on patient anxiety management, effective information provision, and counseling techniques for time-limited day surgery settings.
  Arms: Intervention Group

SUMMARY:
This pilot feasibility study evaluates whether a virtual reality (VR) educational program can help nursing students develop better skills for counseling day surgery patients.

Day surgery patients spend limited time in the hospital but need comprehensive information about their surgery, recovery, and self-care at home. Nurses must provide effective patient education within short timeframes, which creates unique challenges. Research shows that surgical patients consistently report needing more education than they currently receive, particularly about managing pain, recognizing complications, and knowing what to expect during recovery.

Traditional nursing education often lacks the patient's perspective and emotional context that characterize real clinical situations. Virtual reality simulation can address this gap by letting nursing students experience healthcare scenarios from the patient's viewpoint in a safe learning environment.

The CINDY (Counseling Intervention for Day Surgery) intervention uses 360-degree VR videos showing day surgery situations from the patient's perspective. Students can practice counseling skills and learn to understand patient concerns before working with actual patients.

This pilot feasibility study will include 60 nursing students from Seinäjoki University of Applied Sciences. Thirty students will receive the CINDY VR intervention alongside their regular education, while 30 students will receive only standard education. The study will run for approximately 6-7 months.

The primary goal is to test whether this VR approach is feasible and acceptable for nursing education. The study will measure:

* How successfully students can be recruited and retained
* Whether students complete the VR program as designed
* Student and educator satisfaction with the learning method
* Technical performance and usability of the VR platform
* Preliminary changes in student counseling competencies

Results will inform the design of a larger study to definitively test whether VR training improves nursing students' patient counseling skills. This research may help nursing programs better prepare students to provide high-quality patient education in day surgery settings.

DETAILED DESCRIPTION:
BACKGROUND AND FRAMEWORK

The CINDY (Counseling Intervention for Day Surgery) educational intervention was systematically developed using the Medical Research Council (MRC) framework for complex intervention development. The intervention addresses the recognized gap in nursing education regarding patient counseling competencies for day surgery settings, where reduced contact time requires highly effective communication skills.

INTERVENTION DEVELOPMENT (MRC PHASE 1)

Following MRC Phase 1 guidelines, the intervention was co-designed through multidisciplinary collaboration with nursing educators, day surgery nurses, and nursing students. Stakeholder evaluation was conducted with nursing educators (n=6-8), day surgery nurses (n=6-8), and graduating nursing students (n=6-8), demonstrating excellent usability with a Post-System Usability Scale (P-SUS) score of 95.0/100 (scores ≥70 indicate good to excellent usability). Phase 1 results will be reported separately.

CURRENT STUDY (MRC PHASE 2)

This pilot feasibility study represents MRC Phase 2 (Feasibility and Piloting) and follows CONSORT extension guidelines for pilot and feasibility trials. The intervention is described according to the TIDieR (Template for Intervention Description and Replication) checklist to ensure comprehensive and replicable reporting.

STUDY DESIGN

This is a non-randomized pilot feasibility study employing a convergent mixed methods approach with parallel groups (intervention n=30, control n=30). The quasi-experimental design compares students receiving the CINDY VR intervention alongside standard perioperative nursing education with students receiving only standard education.

INTERVENTION DESCRIPTION

The CINDY intervention is a 90-minute VR-based educational program delivered through the ThingLink platform. The intervention was developed through a co-design process involving the principal investigator (nursing educator), a digital content expert, and an experienced day surgery nurse, ensuring both pedagogical soundness and clinical authenticity.

Students experience interactive 360-degree VR scenarios depicting day surgery patient journeys from admission through discharge, including preoperative preparation, postoperative recovery, and discharge counseling. The scenarios were filmed in authentic clinical settings and feature real patient perspectives and concerns. The intervention emphasizes patient perspective-taking, anxiety management strategies, and effective information provision techniques tailored to the time constraints of day surgery settings.

DATA COLLECTION

Mixed methods data collection occurs at three timepoints: baseline (T1), immediately post-intervention (T2), and 4-6 weeks post-intervention (T3). Quantitative measures include patient counseling competencies (OKO Scale), system usability (Post-System Usability Scale), and feasibility indicators (recruitment, retention, adherence, fidelity, acceptability). Qualitative data include semi-structured interviews with students, educators, and day surgery nurses. Intervention group focus group discussions use the TIDieR checklist components as a framework to systematically evaluate intervention delivery, materials, procedures, and fidelity.

PRIMARY OUTCOMES

As a pilot feasibility study, primary outcomes focus on feasibility indicators: recruitment success (≥70% eligible students enrolled), retention (≥80% complete all measurements), intervention adherence (≥75% complete full VR program), intervention fidelity (≥85% scenarios completed correctly), and acceptability (mean P-SUS score ≥70). These predetermined success criteria will inform decisions about proceeding to a definitive randomized controlled trial.

ETHICAL CONSIDERATIONS

The study received ethics approval from Seinäjoki University of Applied Sciences Ethics Committee. All participants provide written informed consent after receiving comprehensive study information. Participation is voluntary with the right to withdraw at any time without consequences to academic standing. Data are managed according to GDPR and Finnish data protection regulations.

SIGNIFICANCE

Results will inform the design and implementation of a future definitive trial to test intervention effectiveness. This research contributes to the evidence base for VR simulation in nursing education and addresses the urgent need for improved patient counseling training in day surgery settings.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in perioperative nursing course at Seinäjoki University of Applied Sciences
* Provided written informed consent
* Basic digital literacy and ability to use computer/tablet devices
* Access to required technology (computer, tablet, or smartphone with internet connection)
* Willingness to participate in all study procedures including surveys and potential interviews

Exclusion Criteria:

* Significant visual or hearing impairments that would prevent use of virtual reality technology
* History of motion sickness or documented intolerance to virtual reality environments
* Current or planned leave of absence during the study period that would prevent completion of all measurement timepoints
* Previous participation in CINDY intervention stakeholder evaluation (Phase 1)
* Inability to read and understand Finnish language study materials

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-11-18 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility Indicators Composite | Baseline to 6-week follow-up
  Composite measure of five feasibility indicators with pre-specified success criteria: (1) Recruitment success: ≥70% of eligible students enrolled; (2) Retention: ≥80% of enrolled students complete all three measurement timepoints; (3) Intervention adherence: ≥75% of intervention group students complete the full 90-minute VR program; (4) Intervention fidelity: ≥85% of VR scenarios completed correctly according to protocol; (5) Acceptability: mean Post-System Usability Scale (P-SUS) score ≥70 among intervention group students. Success defined as meeting at least 4 of 5 pre-specified criteria.

SECONDARY OUTCOMES:
Patient Counselling Competencies | Baseline (T1), immediately post-intervention (T2), and 4-6 weeks post-intervention (T3)
  Measured using the OKO Scale (Ohjausosaamisen kehittymisen seuranta - Patient Counseling Competency Development Assessment Scale), a validated self-assessment instrument evaluating nursing students' patient counseling competencies across multiple domains including communication skills, patient education, and counseling techniques. The OKO Scale consists of 42 items scored on a numeric scale ranging from 0 to 10, where 0 indicates very poor competence and 10 indicates very high competence. Higher scores indicate better patient counseling competency.
Qualitative User Experience | Post-intervention period, within 4-6 weeks after intervention completion
  Semi-structured interviews and focus group discussions exploring students', educators', and day surgery nurses' experiences with the CINDY intervention, including perceived benefits, challenges, suggestions for improvement, and insights into intervention mechanisms. Intervention group students participate in focus groups using TIDieR checklist components as framework.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect student privacy and comply with GDPR and Finnish data protection regulations. Aggregated, de-identified results will be published in peer-reviewed journals and presented at conferences.

REFERENCES:
- [Result] Hoffmann TC, Glasziou PP, Boutron I, Milne R, Perera R, Moher D, Altman DG, Barbour V, Macdonald H, Johnston M, Lamb SE, Dixon-Woods M, McCulloch P, Wyatt JC, Chan AW, Michie S. Better reporting of interventions: template for intervention description and replication (TIDieR) checklist and guide. BMJ. 2014 Mar 7;348:g1687. doi: 10.1136/bmj.g1687. PMID 24609605
- [Result] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Result] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223